CLINICAL TRIAL: NCT01084278
Title: Single-Dose, Open-Label Study of the Pharmacokinetics, Safety, and Tolerability of Colcrys (Colchicine, USP) Tablets 0.6 mg Administered to Healthy Subjects and Subjects With Mild, Moderate, Severe Renal Impairment, and End-Stage Renal Disease
Brief Title: Healthy and Renal Impairment Study of Colcrys (Colchicine, USP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-09-1028; U1111-1132-3386 (Registry Identifier: WHO)
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-09

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Healthy (Experimental): Healthy participants with normal renal function (Creatinine Clearance [CrCl] ≥90 mL/min) received one colchicine 0.6 mg tablet on study day 1.
  Interventions: Drug: Colchicine
- Mild renal impairment (Experimental): Participants with mild renal impairment (estimated Glomerular Filtration Rate [eGFR] 60 to 89 mL/min) received one colchicine 0.6 mg tablet on study day 1.
  Interventions: Drug: Colchicine
- Moderate renal impairment (Experimental): Participants with moderate renal impairment (CrCl/eGFR 30 to 59 mL/min) received one colchicine 0.6 mg tablet on study day 1.
  Interventions: Drug: Colchicine
- Severe renal impairment (Experimental): Participants with severe renal impairment (eGFR 15 to 29 mL/min) received one colchicine 0.6 mg tablet on study day 1.
  Interventions: Drug: Colchicine
- End stage renal disease (ESRD) (Experimental): Participants with end stage renal disease (ESRD) received one colchicine 0.6 mg tablet on study day 1 immediately following dialysis. After a 14-day washout, participants received one colchicine 0.6 mg tablet on Day 15 prior to dialysis.
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — Colchicine tablets
  Other Names: COLCRYS

SUMMARY:
The primary objective of this study is to compare the pharmacokinetic profiles of colchicine and its primary metabolites in plasma and urine following a single 0.6 mg oral dose of colchicine in healthy adults with normal renal function, in patients with mild, moderate or severe renal impairment, and in patients with end-stage renal disease on hemodialysis. An additional objective of this study is to study the clearance of colchicine and its metabolites by hemodialysis. Secondary objectives include evaluation of the safety and tolerability of colchicine in the study population.

DETAILED DESCRIPTION:
40 male and female subjects will be enrolled in the study and stratified into one of five groups based on their renal status as determined from creatinine clearance (CrCL) estimated using the serum creatinine (sCR) and the Cockcroft-Gault and Modified Diet in Renal Disease (MDRD) equations as follows: Treatment group 1 - healthy adults with normal renal function (CrCL/eGFR> 90 mL/min); Treatment groups 2, 3 and 4 - patients with mild (CrCL/eGFR 60-89 mL/min), moderate (CrCL/eGFR 30 to 59 mL/min), and severe (CrCL/eGFR 15 to 29 mL/min) renal impairment, respectively; and Treatment group 5 - subjects with end-stage renal disease requiring hemodialysis. On study day 1, participants in Treatment Groups 1 to 4 will be administered one colchicine 0.6 mg tablet at 8 a.m. under standard fasting conditions. Blood samples will be collected from all participants before dosing and both blood and urine samples will be collected for 120 hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of colchicine and its primary metabolites. There will be two study periods for treatment group 5; Period 1 off dialysis and Period 2 on dialysis with a 14 day washout period between the two study periods. On study day 1, participants in treatment group 5 will be administered one colchicine 0.6 mg tablet under standard fasting conditions immediately following dialysis. Blood samples will be collected from all participants before dosing and for up to 70 hours post-dose at times sufficient to adequately determine the pharmacokinetics of colchicine and its primary metabolites. All adverse events will be evaluated by the investigator and reported in the participant's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females 18-70 years old with a body mass index of <39 kg/m^2.
* Patients with normal renal function or mild renal impairment should be generally healthy on the basis of medical history and physical exam.
* Patients with moderate to end stage renal impairment should be generally medically healthy other than with respect to the morbidities associated with impaired renal function.
* Non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures).

Exclusion Criteria:

* Known hypersensitivity to colchicine or any component of the formulation of the study drug.
* Patients with a history or presence of a significant medical condition that would interfere with interpretation of the study results.
* Patients who have used any drugs or substances known to inhibit or induce cytochrome P450 (CYP) enzymes and/or P-glycoprotein within 28 days prior to the first dose and throughout the study.
* Patients with recent (2 year) history or evidence of alcoholism or drug abuse or significant psychiatric disease.
* Patients with chronic hepatic dysfunction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, MD, Study Chair — Mutual Pharmaceutical Company, Inc.; Javier T Quesada, DO, Principal Investigator — West Coast Clinical Trials, LLC
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at three investigative sites in the United States from 25 May 2010 to 28 February 2011.
Pre-assignment Details: Healthy participants, participants with mild, moderate or severe renal impairment and participants with end stage renal disease (requiring hemodialysis) were stratified to one of five treatment groups based on their renal status. All participants received 0.6 mg colchicine.
Groups:
- Mild: Participants with mild renal impairment (estimated Glomerular Filtration Rate [eGFR] 60 to 89 mL/min) received one colchicine 0.6 mg tablet on study day 1.
- Moderate: Participants with moderate renal impairment CrCl/eGFR 30 to 59 mL/min) received one colchicine 0.6 mg tablet on study day 1.
- Severe: Participants with severe renal impairment (eGFR 15 to 29 mL/min) received one colchicine 0.6 mg tablet on study day 1.
- ESRD: Participants with end stage renal disease (ESRD) received one colchicine 0.6 mg tablet on study day 1 immediately following dialysis. After a 14-day washout, participants received one colchicine 0.6 mg tablet on Day 15 prior to dialysis.
Period: Overall Study
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD
Started | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 52.5 (5.29) | 63.9 (3.94) | 63.0 (5.4) | 57.6 (8.48) | 42.2 (12.85) | 55.85 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 4 | 4 | 20
  Male | 4 | 4 | 4 | 4 | 4 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 0 | 0 | 2
  Black or African American | 0 | 0 | 3 | 3 | 6 | 12
  Native Hawaiian or other pacific islander | 0 | 0 | 0 | 0 | 0 | 0
  White | 8 | 6 | 4 | 4 | 2 | 24
  Other | 0 | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 5 | 3 | 3 | 1 | 0 | 12
  Not Hispanic or Latino | 3 | 5 | 5 | 7 | 8 | 28
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 8 | 40
Child Bearing Potential [Number; unit: participants] — Counts are based on the number of female participants.
  participants
    Yes | 0 | 0 | 1 | 0 | 2 | 3
    No | 4 | 4 | 3 | 4 | 2 | 17
Creatinine Clearance/estimated Glomerular Filtration Rate [Mean (Standard Deviation); unit: mL/min] — Creatinine Clearance for Healthy Treatment Group and estimated Glomerular Filtration Rate for Mild, Moderate, Severe and ESRD Treatment Groups.
  mL/min | 111.49 (22.651) | 73.3 (8.10) | 40.0 (6.78) | 22 (4.17) | 10.9 (2.97) | 55.70 (36.61)
Height [Mean (Standard Deviation); unit: cm] | 170.33 (7.722) | 167.94 (8.865) | 164.83 (9.054) | 172.06 (8.643) | 168.05 (11.991) | 169.09 (9.27)
Weight [Mean (Standard Deviation); unit: kg] | 77.09 (8.494) | 65.55 (9.904) | 77.55 (10.667) | 100.81 (16.856) | 73.86 (22.287) | 78.95 (18.47)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.54 (2.113) | 23.18 (2.560) | 28.64 (4.823) | 33.96 (4.489) | 25.66 (5.018) | 27.60 (5.28)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration of colchicine in the plasma.
Time Frame: Day 1 and Day 15 (for ESRD patients only) pre-dose and at 0.5, 1, 1.5 , 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 hours post dose
Population: Per Protocol Analysis Population - Participants renal function was characterized by CrCl using the Cockcroft-Gault equation as healthy (≥90 mL/min), and characterized by Modified Diet in Renal Disease (MDRD) equations as mild (60 - 89 mL/min), moderate (30 - 59 mL/min), severe (15 - 29 mL/min), and ESRD patients requiring dialysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Healthy: Healthy participants with normal renal function received one colchicine 0.6 mg tablet on study day 1.
- Mild: Participants with mild renal impairment received one colchicine 0.6 mg tablet on study day 1.
- Moderate: Participants with moderate renal impairment received one colchicine 0.6 mg tablet on study day 1.
- Severe: Participants with severe renal impairment received one colchicine 0.6 mg tablet on study day 1.
- ESRD - Off Dialysis: Participants with end stage renal disease (ESRD) received one colchicine 0.6 mg tablet taken on study day 1 immediately following dialysis.
- ESRD - on Dialysis: Participants with end stage renal disease (ESRD) received one colchicine 0.6 mg tablet on Day 15 prior to dialysis.
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD - Off Dialysis | ESRD - on Dialysis
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
ng/mL | 2.43 (0.68) | 2.73 (0.78) | 3.69 (1.42) | 2.53 (0.73) | 2.67 (0.94) | 2.27 (0.71)

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: The time to reach the maximum or peak concentration of colchicine in the plasma.
Time Frame: Day 1 and Day 15 (for ESRD patients only) at 0.5, 1, 1.5 , 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD - Off Dialysis | ESRD - on Dialysis
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
hours | 1.31 (0.37) | 1.01 (0.04) | 1.31 (0.37) | 1.58 (0.68) | 1.31 (0.46) | 1.29 (1.01)

3. Primary Outcome: Area Under the Concentration Time Curve From Time Zero to the Time of Last Measured Concentration (AUC 0-t)
Description: The area under the plasma concentration versus time curve beginning from the first dose until the last quantifiable concentration, calculated by the linear trapezoidal method.
Time Frame: Day 1 and Day 15 (ESRD patients only), predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD - Off Dialysis | ESRD - on Dialysis
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
ng*h/mL | 23.37 (7.75) | 25.83 (5.43) | 43.94 (11.68) | 40.44 (13.58) | 26.09 (8.73) | 22.65 (8.54)

4. Primary Outcome: Area Under the Concentration Time Curve From Time Zero to Infinity (AUC 0 - ∞)
Description: The area under the plasma concentration versus time curve extrapolated to infinity. AUC 0 - ∞ is calculated as the sum of total AUC 0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD - Off Dialysis | ESRD - on Dialysis
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
ng*h/mL | 24.73 (8.10) | 27.21 (5.56) | 48.94 (13.45) | 48.00 (17.36) | 31.68 (12.28) | 30.61 (17.29)

5. Primary Outcome: Apparent First-order Terminal Elimination Rate Constant (Kel)
Description: Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma concentration versus time curve for colchicine. The parameter was calculated by linear least-squares regression analysis using the maximum number of points in the terminal log-linear phase (e.g., three or more non-zero plasma concentrations).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD - Off Dialysis | ESRD - on Dialysis
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
1/hr | 0.023 (0.004) | 0.023 (0.003) | 0.018 (0.002) | 0.014 (0.002) | 0.025 (0.006) | 0.020 (0.007)

6. Primary Outcome: Apparent First-order Terminal Elimination Half-life (t½)
Description: The apparent first-order terminal elimination half-life was calculated as 0.693/Kel.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD - Off Dialysis | ESRD - on Dialysis
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
hr | 30.63 (5.43) | 30.92 (3.54) | 39.90 (3.93) | 49.53 (6.01) | 29.38 (7.51) | 40.80 (21.71)

7. Primary Outcome: The Apparent Total Volume of Distribution After Administration (V-area/F)
Description: The apparent total volume of distribution after administration of colchicine, calculated as Dose / (AUC0-∞ × Kel).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD - Off Dialysis | ESRD - on Dialysis
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
L | 1131.68 (247.32) | 1024.22 (266.47) | 761.81 (237.07) | 1009.02 (419.88) | 870.46 (230.68) | 1263.0 (462.40)

8. Primary Outcome: Weight-adjusted Apparent Total Volume of Distribution After Administration (V-area/F)
Description: The apparent total volume of distribution after administration of colchicine, calculated as Dose / (AUC0-∞ × Kel), and normalized to body weight.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD - Off Dialysis | ESRD - on Dialysis
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
L/kg | 14.84 (3.36) | 15.80 (3.94) | 10.06 (3.65) | 9.91 (3.10) | 13.35 (6.94) | 18.91 (11.91)

9. Primary Outcome: Apparent Total Body Clearance of Colchicine
Description: The apparent total body clearance after administration of colchicine, calculated as Dose/AUC(0-∞).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD - Off Dialysis | ESRD - on Dialysis
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
L/hr | 26.34 (7.57) | 23.04 (5.60) | 13.63 (5.80) | 14.59 (7.37) | 22.07 (9.87) | 25.78 (15.08)

10. Primary Outcome: Weight-adjusted Apparent Total Body Clearance of Colchicine
Description: The apparent total body clearance after administration of colchicine, calculated as Dose/AUC(0-∞) and normalized to body weight (in kilograms).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr/kg
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD - Off Dialysis | ESRD - on Dialysis
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
L/hr/kg | 0.34 (0.08) | 0.36 (0.12) | 0.18 (0.09) | 0.14 (0.06) | 0.35 (0.26) | 0.41 (0.36)

11. Primary Outcome: Amount of Colchicine Excreted in Urine (Ae[0-t])
Description: The amount of colchicine excreted in urine during the post-dose collection, calculated as the sum of the amounts in the individual collection intervals (Ae).
Time Frame: Pre-dose on Day 1 and up to 120 hours post dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 8 | 8 | 8 | 8
mg | 0.110 (0.032) | 0.100 (0.026) | 0.094 (0.053) | 0.058 (0.012)

12. Primary Outcome: Percentage of Colchicine Dose Excreted in Urine up to the Final Collection Time
Description: The cumulative percentage of the colchicine dose excreted in urine up to the final collection time, calculated as Ae(0-t) × 100/dose
Time Frame: Pre-dose on Day 1 and up to 120 hours post dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of dose
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 8 | 8 | 8 | 8
percent of dose | 18.34 (5.39) | 16.69 (4.3) | 15.67 (8.77) | 9.63 (2.05)

13. Primary Outcome: Renal Clearance of Colchicine (CLR)
Description: Renal clearance of colchicine, calculated as Ae(0 t)/AUC 0-t.
Time Frame: Pre-dose on Day 1 and up to 120 hours post dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 8 | 8 | 8 | 8
L/hr | 4.78 (0.51) | 3.90 (0.74) | 2.12 (0.86) | 1.69 (1.13)

14. Primary Outcome: Dialysis Clearance of Colchicine (CLD)
Description: The dialysis clearance of colchicine, calculated as amount of colchicine recovered in dialysate / AUCt2-t1 where t1 and t2 are the times of the start and end of hemodialysis.
Time Frame: Day 15, post-dose during dialysis
Population: ESRD participants on dialysis, where data were available.
Measure: Mean (Standard Deviation); unit: L/h
Groups:
- End Stage Renal Disease (ESRD): Participants with end stage renal disease (ESRD) received one colchicine 0.6 mg tablet taken under standard fasting conditions on study day 1 immediately following dialysis. After a 14-day washout, participants received one colchicine 0.6 mg tablet on Day 15 prior to dialysis.
Arm/Group | End Stage Renal Disease (ESRD)
Number analyzed (Participants) | 7
L/h | 7.4 (0.7)

15. Primary Outcome: Percentage of Colchicine Dose Recovered in Dialysate
Description: The cumulative percentage of the colchicine dose recovered in dialysate.
Time Frame: Day 15, post-dose during dialysis
Population: ESRD participants on dialysis, where data were available.
Measure: Mean (Standard Deviation); unit: percent dose
Arm/Group | End Stage Renal Disease (ESRD)
Number analyzed (Participants) | 7
percent dose | 5.2 (2.3)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 6 days.
Description: The investigator documented any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Healthy | Mild | Moderate | Severe | ESRD
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 2/8 | 4/8 | 4/8 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy (N=8) | Mild (N=8) | Moderate (N=8) | Severe (N=8) | ESRD (N=8)
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1
Infusion site erythema (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion site induration (General disorders) | 0 | 0 | 0 | 1 | 0
Medical device complication (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 2 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.